CLINICAL TRIAL: NCT02381223
Title: Simplified Medical Abortion Screening: A Pilot Demonstration Project
Status: Completed | Type: Observational
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Other Study IDs: 1020
Record Dates: First submitted 2015-02-23; First posted 2015-03-06 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Medical; Abortion, Fetus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to collection additional data on the safety and acceptability of medical abortion without pretreatment pelvic ultrasound or exam in woman who meet certain criteria.

ELIGIBILITY:
Inclusion criteria:

* Women having medical abortion

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Female: only female participants are being studied
Sampling Method: Non-Probability Sample
Enrollment: 409 (Actual)
Dates: Start 2015-03; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse events | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Raymond, MD, Principal Investigator — Gynuity Health Projects
Locations (5):
- United States (3):
  - Carafem, Friendship Heights, Maryland
  - Planned Parenthood Minnesota, North Dakota, South Dakora, Minneapolis, Minnesota
  - Institute for Family Health, New York, New York
- Centro de Salud Mexico-Espana, Mexico City, Mexico
- Reproductive Health Training Center, Chisinau, Moldova

REFERENCES:
- [Derived] Raymond EG, Tan YL, Comendant R, Sagaidac I, Hodorogea S, Grant M, Sanhueza P, Van Pratt E, Gillespie G, Boraas C, Weaver MA, Platais I, Bousieguez M, Winikoff B. Simplified medical abortion screening: a demonstration project. Contraception. 2018 Apr;97(4):292-296. doi: 10.1016/j.contraception.2017.11.005. Epub 2017 Nov 21. PMID 29170088